CLINICAL TRIAL: NCT07381790
Title: Modern Technologies for Individual Risk Stratification in Infant Lower Respiratory Tract Infections
Brief Title: Modern Technologies in Lower Respiratory Tract Infections in Children
Acronym: MoT-LRTI
Status: Recruiting | Type: Observational
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 940358
Record Dates: First submitted 2025-12-02; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Bronchiolitis Acute; Lower Respiratory Tract and Lung Infections; Pediatric Lung Ultrasound; Tidal Volume; Pediatric Lung Diagnosis; Pediatric Asthma
Keywords: pediatric; lung ultrasound; lower respiratory tract infections; tidal-flow volume loops

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- children under 2 years of age, hospitalized with lower respiratory tract infection
  Interventions: Diagnostic Test: lung ultrasound; Diagnostic Test: Tidal-flow volume loops

INTERVENTIONS:
Diagnostic Test: lung ultrasound — performance of lung utltrasound in participants, performed bedside (v scan).
Diagnostic Test: Tidal-flow volume loops — tidal-flow volume loops performed in patients hospitalized with lower respiratory tract infections.

SUMMARY:
Lower respiratory tract infections (LRTIs) are a significant cause of childhood morbidity and mortality globally, particularly in low-income countries. In Norway, LRTIs is a leading cause of hospitalization among infants, representing a great socioeconomic burden.

Bronchiolitis, a viral infection, is the main representation of LRTIs in infants. It affects the small airways, causing breathing- and feeding difficulties. Today, treatment relies on subjective evaluations, lacking objective measures for assessment. This increases the risk of both under- and over treating patients. In the long term, bronchiolitis increases risk of asthma, but it is unknown who the high-risk patients for chronic lung disease are.

Lung ultrasonography (LUS) has emerged as a promising tool for assessing bronchiolitis severity and progression of the disease. The investigators will explore its use to improve diagnostic accuracy and treatment decisions, and develop AI-driven scoring tools for novel technology.

Additionally, tidal breathing flow volume loops (TBFVL) offer a non-invasive method for evaluating airway obstruction in infants, with the potential to assess severity of bronchiolitis, treatment efficacy and post-infection lung function.

In this project the investigators will combine the use of these modern technologies to improve treatment and follow-up of infants with LRTIs.

The main aim for this observational study is to assess the utility of lung ultrasonography (LUS) and tidal flow volume loops (TBFVL) in infant lower respiratory tract infections (LRTIs) for individual risk stratification in acute and chronic settings. This aims to refine the management of bronchiolitis, identifying high-risk patients for chronic lung disease to tailor treatment and follow-up protocols.

The project has three secondary objectives.

1. To assess correlation between LUS and TBFVL findings with clinical score at admission, length of stay, need of respiratory support and ICU admissions.
2. To assess duration of symptoms following acute bronchiolitis and evaluate the use of LUS and TBFVL in objectively examine post-infectious sequela.
3. To evaluate the long-term impact of bronchiolitis on lung function through clinical follow-up after a 12 month period.

Lower respiratory tract infections (LRTIs) stand as the leading cause of hospitalization, while asthma is the leading cause of chronic lung disease among children in Nordic countries. The project seeks to improve risk stratification and treatment protocols in both acute and chronic settings.

In the acute setting, the project endeavors to prognosticate individual patient outcomes, thereby individualize treatment and mitigating unnecessary hospital admissions, use of respiratory support and antibiotic administration. Additionally there is potential of more aggressive treatment to selected patients. The study aims to improve the understanding of pathophysiological processes of LRTIs in infants, providing objective metrics to evaluate disease severity and individualize treatment.

The investigators aim to validate the utility, validity, and simplicity of handheld ultrasound devices as bedside diagnostic tools for this common disease, alongside affirming the value of tidal flow volume loops (TBFVL) in acute and chronic settings to assess airway obstruction in infants. Combining these modern technologies, evaluating affliction of both the parenchyme and the airways will probide a new perspective in treatment of LRTIs. In addition the project will strive to develop novel technology with AI-driven scoring tools of LUS.

Furthermore, the project aims to examine the trajectory of symptoms post-LRTI and facilitate the early identification of patients with high-risk of chronic lung disease. Early detection of asthma and other chronic lung diseases holds the potential to improve outcomes and mitigate the need for hospitalization, thus easing both economic and emotional burdens associated with the disease.

For caregivers, the lack of information concerning symptom duration and risk of future disease represents a significant knowledge gap. The project aims to address this, by examining post-infection symptom duration and identifying high-risk cohorts predisposed to chronic lung disease. This has the potential to both improve information, personalize follow-up and reduce hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of lower respiratory tract infection
* with tachypnea and/or
* wheezing
* Retractions
* Respiratory difficulties

Exclusion Criteria:

* Severe Congenital heart disease (not ASD, small VSD, PDA)
* Cystic fibrosis and PCD
* Neuromuscular diseases and other diseases with reduced airway clearance
* Severe malacia, diagnosed by bronchoscopy by time of T0.
* Foreign body inhalation
* Pneumothorax
* Pleural effusion (with need of invasive interventions)
* Bronchopulmonary dysplasia or GA <32 weeks
* Caretaker not able to communicate in Norwegian or English
* Weight <3 kg

Ages: 0 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children under 2 years of age, hospitalized with lower respiratory tract infections. single cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of readmissions at 1 year follow-up after baseline. | From enrollment to the end of follow-up at 12 months.
  All participants will be followed for 1 year after first hospitalization with LRTI. At that point investigators will retrieve data on readmissions as primary outcome, correlated with initial findings.
Length of stay at hospital due to LRTI. | from enrollment to discharge from hospital, average patient is hospitalized 3 days.
  Primay outcome is length of stay at hospital, correlated with findings at hospitalization (lung ultrasound and tidal-flow volume loops)
Duration of symptoms after hospitalization due to LRTI. | from enrollment to weeks/months after discharge, based on reporting of symptoms. Up to 60 days.
  duration of symptoms after hospitalization with lower respiratory tract infection, marked by symptom diary and follow-up by phone call. Participants are deemed free of symptoms when they are in habitual state without cough.

SECONDARY OUTCOMES:
Use of respiratory support correlated with lung ultrasound score and tidal-flow volume loop results | form enrollment to discharge from hospital, average hospitalization is 3 days.
  secondary outcome is degree of respiratory support correlated with findings on lung ultrasound (LUS) and tidal-flow volume loops (TBFVL). Investigators will monitor the use of NIV (HFNC, C-PAP, mechanical ventilation) in enrolled participants and correlate with results from TBFVL and scoring from LUS.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Aalesund Hospital, Ålesund, Møre og Romsdal
  - St. Olavs Hospital HF, Trondheim, Sør-Trøndelag

IPD SHARING:
Plan to Share IPD: No